CLINICAL TRIAL: NCT00524212
Title: Ph. D Student, Jane Byriel Knudsen, Aarhus University
Brief Title: How to Improve Diagnosis in Infective Endocarditis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Jane Byriel Knudsen, Dept. of Cardiology, Aarhus University Hospital, Skejby - Denmark
Other Study IDs: 06-10-B640-A1205-22345; 20060181; SUN-2007-653
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Endocarditis, Bacterial
MeSH Terms: conditions — Endocarditis, Bacterial

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A venous blood sample was obtained from each patients and all samples were centrifuged and immediately frozen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IE confirmed IE rejected: Prospective, controlled, blinded study of clinical/TEE criteria of IE compare to clinical/blood test criteria of IE.
- IE confirmed IE rejected

SUMMARY:
The purpose is to exam prospective if simple clinical information in combination with a normal s-procalcitonin are sufficient for exclusion of infective endocarditis (IE).

DETAILED DESCRIPTION:
Despite progress in surgical and medical treatment, infective endocarditis is still associated with high morbidity and mortality.

The variable clinical presentation of IE makes the diagnosis a clinical challenge.

Procalcitonin is a precursor from the hormone calcitonin and also a marker of systemic bacterial infections.

The purpose of this study is:

* to investigate the diagnostic value of serum procalcitonin (PCT), C-reactive protein (CRP) and sedimentation rate (SR) when IE is suspected.
* to investigate if a retrospectively generated clinical model suitable for exclusion of IE can be confirmed prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 18 year with suspected or verified Infective Endocarditis
* By word of mouth or in writing consent

Exclusion Criteria:

* Incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort was selected from all the patients admitted to the tertiary hospital (the initial diagnosis was infective endocarditis)
Sampling Method: Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2007-03; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane B Knudsen, Dr., Principal Investigator — Aarhus University Hospital, Skejby, Department of Cardiology, 8200 Aarhus N, Denmark
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus, Denmark